CLINICAL TRIAL: NCT00378534
Title: Peripheral Blood Stem Cell Allotransplantation for Hematological Malignancies Using a Positive Stem Cell Selection Technique for T Cell Depletion, Followed by Delayed T Cell Add-Back
Brief Title: Methods to Enhance the Safety and Effectiveness of Stem Cell Transplants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060248; 06-H-0248 (Other: NIH National Heart, Lung and Blood Institute); NCT00398346 (obsolete NCT alias)
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2014-12

CONDITIONS: Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: Chronic Myelogenous Leukemia (CML); Acute Myelogenous Leukemia (AML); Chronic Lymphocytic Leukemia (CLL); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS); Leukemia; Chronic Myelogenous Leukemia; CML; Acute Myeloid Leukemia; AML; Chronic Lymphocytic Leukemia; CLL; Acute Lymphoblastic Leukemia; ALL; Myelodysplasia Syndrome
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia | interventions — fludarabine; fludarabine phosphate; Cyclosporine; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T Cell Depletion Transplant Participants (Experimental): Participants with hematological malignancies received a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation followed by an infusion of stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a delayed T cell depletion add back as donor lymphocyte infusion at day 90.
  Interventions: Device: Miltenyi reagent system; Drug: Fludarabine; Drug: Cyclosporine; Drug: Cyclophosphamide
- Stem Cell Donors (Other): An HLA 6/6 identical family member will be co-enrolled into this study as a stem cell donor. The stem cell collection aspect of this protocol is not investigational.
  Interventions: Other: FILGRASTIM (G-CSF)

INTERVENTIONS:
Device: Miltenyi reagent system — Miltenyi Clinimax CD34 Reagent System for CD34 selection and delayed T cell depletion add back
  Other Names: Miltenyi Clinimax CD34 Reagent System
  Arms: T Cell Depletion Transplant Participants
Drug: Fludarabine — Therapeutic
  Other Names: Fludara
  Arms: T Cell Depletion Transplant Participants
Drug: Cyclosporine — Therapeutic
  Other Names: Neoral
  Arms: T Cell Depletion Transplant Participants
Drug: Cyclophosphamide — Therapeutic
  Other Names: Cytoxan
  Arms: T Cell Depletion Transplant Participants
Other: FILGRASTIM (G-CSF) — An HLA 6/6 identical family member will be co-enrolled into this study as a stem cell donor. Stem cell Donors will receive G-CSF for stem cell mobilization. The stem cell collection aspect of this protocol is not investigational.
  Other Names: Neupogen
  Arms: Stem Cell Donors

SUMMARY:
Bone marrow stem cell transplants (otherwise called bone marrow transplants) from healthy donors are sometimes the only means of curing hematological malignant diseases such as acute and chronic leukemias, myelodysplastic syndrome, myeloproliferative diseases and lymphomas. Before transplant the patient receives chemotherapy and radiation treatment to reduce the malignancy to low levels and to prevent rejection of the transplant. The transplant restores the blood counts to normal and replaces the patients immunity with that of the donor. The donors immune cells increase the effect of the transplant by attacking remaining malignant cells. Donor immune cells (especially those called T lymphocytes) also attack healthy non-cancerous cells and tissues of the recipient causing "graft-versus-host-disease" (GVHD). Strong GVHD reactions occurring within weeks after the transplant can be life-threatening . In this study we remove most of the T lymphocytes from the transplant to minimize the risk of GVHD. However to improve immunity against residual malignant cells and boost immunity to infections, donor T cells (stored frozen at time of transplant) are given back around 90 days after the transplant when they have a reduced risk of causing serious GVHD.

Any patient between 10 and 75 years of age with acute or chronic leukemia, myelodysplastic syndrome, myeloproliferative syndromes or lymphoma, who have a family member who is a suitable stem cell donor may be eligible for this study. Candidates are screened with a medical history and various tests and examinations.

DETAILED DESCRIPTION:
Peripheral blood stem cell transplant research carried out by the National Heart Lung and Blood Institute (NHLBI) Bone Marrow Transplantation (BMT) Unit focus on transplant techniques designed to decrease graft versus host disease (GVHD), increase the graft-versus-leukemia (GVL) effect and reduce the risk of post-transplant graft rejection.

We have found that by controlling the stem cell (CD34+ cell) and T lymphocyte (CD3+ cell) dose severe GVHD can be reduced whilst beneficial GVL effects can be preserved by postponed donor lymphocyte infusion (DLI). We found that T cell depleted transplants using the Nexell/Baxter Isolex 300i system to obtain high CD34+ doses depleted of lymphocytes were safe to administer and associated with less severe acute GVHD and promising response rates and overall survival, when combined with a delayed T cell add-back (DLI). This protocol is designed to evaluate safety and efficacy of an improved T cell depletion procedure using the Miltenyi CliniMACs system (CD34 reagent system) with a delayed T cell add back in the HLA-matched peripheral blood stem cell transplant setting.

The protocol will accrue up to 68 subjects ages 10-75 with a hematological malignancy, in whom allogeneic stem cell transplantation from an HLA-matched sibling would be routinely indicated. 68 sibling donors will also be recruited. Diagnostic categories will include acute and chronic leukemia, myelodysplastic syndrome, lymphoma, multiple myeloma and myeloproliferative syndromes.

Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection, and a delayed T-cell add back as donor lymphocyte infusion (DLI) at day 90. Older subjects will receive a lower dose of irradiation to reduce the regimen intensity.

Participants undergo apheresis to collect lymphocytes for research studies. This procedure involves collecting blood through a needle in the arm, extracting the lymphocytes through a cell separator machine and returning the rest of the blood through a needle in the other arm. Before treatment begins, patients have a central intravenous line (plastic tube) placed in a vein in the neck. This line remains in place during the transplant and recovery period for drawing and transfusing blood, giving medications, and infusing the donated cells.

To prepare patients for transplantation their immune system is suppressed by a combination of chemotherapy and radiation which will also help to fight remaining malignant cells. The chemotherapy consists of two anti-cancer drugs (fludarabine and cyclophosphamide) and will be infused over the central line starting eight days before the transplant. Patients will receive eight doses of total body irradiation, administered in two 30-minute sessions per day for 4 days. Patients above 55 years of age who tolerate transplants less well than younger individuals will receive a lower dose of radiation. One day after the preparative treatment is finished, patients receive the transplant of donors stem cells as an infusion through the central line.

Patients receive cyclosporine, an immunosuppressive drug starting 6 days before the transplant until 21 days post-transplant. This helps prevent both transplant rejection and GVHD. The drug is stopped to allow the donor immunity to function and is restarted on day 89 to prevent GVHD from the infusion of T lymphocytes on day 90.

Patients are followed with various tests, treatments and examinations periodically for the first 3 years and then yearly thereafter.

Primary endpoint will be overall survival at day +200. Non-relapse mortality at day +200 will be monitored for safety. Secondary endpoints will be standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD and relapse of disease.

ELIGIBILITY:
INCLUSION CRITERIA - RECIPIENT:

* Ages 10-75 years inclusive
* Chronic myelogenous leukemia (CML):
* Subjects under the age of 21 in chronic phase
* Subjects ages 10-75 in chronic phase who have failed treatment with imatinib, have intolerance to imatinib, or who did not receive imatinib at therapeutic doses within the first 12 months from diagnosis.
* Subjects ages 10-75 in accelerated phase or blast transformation.
* Acute lymphoblastic leukemia (ALL): any of these categories: ALL in first remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, Karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia) All second or subsequent remissions, primary induction failure, partially responding or untreated relapse.
* Acute myelogenous leukemia (AML): AML in first remission - except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse
* Myelodysplastic syndromes (MDS): any of these categories - refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia, atypical MDS/myeloproliferative syndromes
* Myeloproliferative disorders including atypical (Ph negative) chronic myeloid and neutrophilic leukemias, progressing myelofibrosis, and polycythemia vera, essential thrombocythemia in transformation to acute leukemia or with progressive transfusion requirements or pancytopenia.
* Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000 /microl) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy.
* Non-Hodgkins lymphoma including Mantle cell lymphoma relapsing or refractory to standard of care treatments
* Multiple myeloma, Waldenstrom's macroglobulinemia, unresponsive or relapsed following standard of care treatments.
* HLA identical (6/6) related donor
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: written informed consent from one parent or guardian. Informed oral consent from minors: the process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA - RECIPIENT:

* Estimated probability of surviving less than three months
* Major anticipated illness or organ failure incompatible with survival from transplant
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and making informed consent impossible.
* Positive pregnancy test for women of childbearing age.
* HIV positive
* Diffusion Capacity of Lung for Carbon Monoxide (DLCO) adjusted for ventilation and hemoglobin less than 65 percent predicted
* Left ventricular ejection fraction less than 40 percent
* Aspartate Aminotransferase (AST)/Serum Glutamate Oxaloacetate Transaminase (SGOT) greater than 10 times upper limit of normal (ULN) (CTCAE grade IV v3.0)
* Bilirubin greater than 5 times upper limit of normal (ULN) (CTCAE grade IV v3.0)
* Creatinine greater than 4.5 times upper limit of normal (ULN) (CTCAE grade IV v 3.0)
* Prior allogeneic stem cell transplantation.

INCLUSION CRITERIA - DONOR:

* Related donor, HLA identical (6/6) with recipient
* Weight greater than or equal to 18 kg
* Age greater than or equal to 2 or less than or equal to 80 years old
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA - DONOR:

* Pregnant. Lactating donors permitted provide breast milk is discarded during the days that G-CSF is given
* Unfit to receive filgrastim (G-CSF) and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension)
* Sickling hemoglobinopathies including HbSS, HbAS, HbSC
* HIV positive donors who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II) will be used at the discretion of the investigator following counseling and approval from the recipient
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minocher M Battiwalla, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Appelbaum FR. Haematopoietic cell transplantation as immunotherapy. Nature. 2001 May 17;411(6835):385-9. doi: 10.1038/35077251. PMID 11357147
- [Background] Armitage JO. Bone marrow transplantation. N Engl J Med. 1994 Mar 24;330(12):827-38. doi: 10.1056/NEJM199403243301206. No abstract available. PMID 8114836
- [Background] Balaguer H, Galmes A, Ventayol G, Bargay J, Besalduch J. Splenic rupture after granulocyte-colony-stimulating factor mobilization in a peripheral blood progenitor cell donor. Transfusion. 2004 Aug;44(8):1260-1. doi: 10.1111/j.1537-2995.2004.00413.x. No abstract available. PMID 15265137
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] McIver Z, Melenhorst JJ, Wu C, Grim A, Ito S, Cho I, Hensel N, Battiwalla M, Barrett AJ. Donor lymphocyte count and thymic activity predict lymphocyte recovery and outcomes after matched-sibling hematopoietic stem cell transplant. Haematologica. 2013 Mar;98(3):346-52. doi: 10.3324/haematol.2012.072991. Epub 2012 Oct 12. PMID 23065508
- [Derived] Melenhorst JJ, Tian X, Xu D, Sandler NG, Scheinberg P, Biancotto A, Scheinberg P, McCoy JP Jr, Hensel NF, McIver Z, Douek DC, Barrett AJ. Cytopenia and leukocyte recovery shape cytokine fluctuations after myeloablative allogeneic hematopoietic stem cell transplantation. Haematologica. 2012 Jun;97(6):867-73. doi: 10.3324/haematol.2011.053363. Epub 2011 Dec 1. PMID 22133778
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0248.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T Cell Depletion Transplant Participants | Stem Cell Donors
Started | 58 | 58
Completed | 55 | 58
Not Completed | 3 | 0
Not completed — Participants did not receive transplant | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T Cell Depletion Transplant Participants | Stem Cell Donors | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 27 | 28 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 31 | 61
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 22 | 20 | 42
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Survival and Non-relapse Mortality at Day +200 Using the Miltenyi Reagent System
Description: Subjects with hematological malignancies receiving a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation followed by an infusion of stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a delayed T cell depletion add back as donor lymphocyte infusion at day 90. The subjects receiving allogeneic stem cell transplantation will have stem cell product prepared using Miltenyi CliniMacs system to determine the overall survival and non-relapse mortality at day +200.
Time Frame: Day 200
Measure: Number; unit: participants
Arm/Group | T Cell Depletion Transplant Participants
Number analyzed (Participants) | 55
participants
  Survival at day 200 | 43
  Non-relapse mortality | 4

2. Secondary Outcome: Number of Participants With Relapse of Disease
Description: Number of participants with relapse of disease by day 200
Time Frame: Day 200
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Transplant Participants
Number analyzed (Participants) | 55
Participants | 17

3. Secondary Outcome: Number of Participants Who Developed Acute GVHD Grades I, II, III, IV
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Transplant Participants
Number analyzed (Participants) | 55
Participants
  Acute GVHD, Grade I | 14
  Acute GVHD, Grade II | 16
  Acute GVHD, Grade III | 9
  Acute GVHD, Grade IV | 1

4. Secondary Outcome: Number of Participants Who Developed Limited Chronic GVHD
Description: Number of incidences of participants who developed Limited Chronic Graft vs Host Disease (GVHD).
  Limited disease is characterized by localized skin involvement and/or evidence of hepatic dysfunction.
  Limited disease is associated with a favorable outcome without systemic therapy, while extensive disease patients have an unfavorable outcome.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Transplant Participants
Number analyzed (Participants) | 55
Participants | 8

5. Secondary Outcome: Number of Participants Who Develop Extensive GVHD
Description: Number of participants with extensive, Chronic Graft vs Host Disease (GVHD). Extensive chronic GVHD is defined as GVHD occurring after day 100 that did not meet the definition of limited chronic GVHD.
  Extensive disease presents either with generalized skin involvement, or with localized skin involvement or hepatic dysfunction plus at least one of the following:
  * Liver histology showing chronic progressive hepatitis, bridging necrosis, or cirrhosis
  * Involvement of the eye (Schirmer's test with less than 5 mm wetting) (see "Diagnosis and classification of Sjögren's syndrome")
  * Involvement of minor salivary glands or oral mucosa (as demonstrated on labial or mucosal biopsy specimen)
  * Involvement of any other target organ
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | T Cell Depletion Transplant Participants
Number analyzed (Participants) | 55
Participants | 18

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | T Cell Depletion Transplant Participants | Stem Cell Donors
All-Cause Mortality (participants affected / at risk) | 14/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 14/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T Cell Depletion Transplant Participants (N=58) | Stem Cell Donors (N=58)
Graft failure (Blood and lymphatic system disorders) | 3 (3) | 0
Infection (Infections and infestations) | 7 (7) | 0
GVHD (Immune system disorders) | 4 (4) | 0
Posterior reversible encephalopathy syndrome (Immune system disorders) | 1 (1) | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0
Arrythmia (Cardiac disorders) | 1 (1) | 0
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 — rectal hemorrhage
Microangiopathy Anemia (Blood and lymphatic system disorders) | 1 (1) | 0
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No